CLINICAL TRIAL: NCT05848206
Title: Impact of Formulary Coverage of Entresto (Sacubitril/Valsartan) on Prescription Abandonment/Rejection and Subsequent Treatment and Economic Outcomes in Chronic Heart Failure Patients in the U.S.
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLCZ696BUS34
Record Dates: First submitted 2023-04-27; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Primary LAAD Cohort: Patients with ≥1 SAC/VAL transactions from plans of interest identified in LAAD
- Secondary LAAD Cohort: Patients with SAC/VAL abandonment or rejection identified in LAAD

SUMMARY:
This was a retrospective cohort study utilizing IQVIA open-source pharmacy and medical claims data among patients with a sacubitril/valsartan (SAC/VAL) prescription transaction.

ELIGIBILITY:
Inclusion Criteria:

Primary IQVIA Longitudinal Access and Adjudication Data (LAAD) Cohort (for primary objective)

* Patients with ≥1 transaction for SAC/VAL in LAAD between 01 January 2017 and 30 November 2019 (index period). Date of the 1st SAC/VAL prescription transaction during this period was the index date.
* Patients from the Novartis-provided list of 21 plans and formularies of interest (mapping to LAAD data was based data elements such as plan name, payer name, and pharmacy benefit manager [PBM] name) as of the index date.
* Patients aged ≥18 years on the index date.
* Patients with 12-months of data visibility pre-index.
* Patients with 3-months of data visibility post-index (to allow for final adjudication/abandonment status confirmation).

For comorbidity data only:

* Patients with linkage of LAAD FIA to LAAD Dx by patient ID.
* Patients with ≥2 non-ancillary medical claims ≥30 days apart within the 12 months pre-index period.

Secondary LAAD Cohort (for secondary objective)

* Among patients from the Primary LAAD Cohort remaining in Step 6, patients who abandoned their 1st SAC/VAL prescription or did not receive SAC/VAL due to claim rejection in LAAD between 01 January 2017 and 28 February 2019 (index period). Date of the 1st abandoned/rejected SAC/VAL prescription transaction during this period is the index date.
* Patients aged ≥18 years on the index date.
* Patients with 12-months of data visibility pre-index.
* Patients with 12-months of data visibility post-index.
* For comorbidity data only:
* Patients with linkage of LAAD FIA to LAAD Dx by patient ID.
* Patients with ≥2 non-ancillary medical claims ≥30 days apart within the 12 months pre-index period.

Exclusion Criteria:

* Patients with a SAC/VAL transaction during the 12-month pre-index period.
* Patients with data quality issues (e.g., missing gender).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 251831 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who had SAC/VAL prescriptions filled | Up to 3 months
Percentage of patients who had abandoned (not accepted) SAC/VAL prescriptions | Up to 3 months
Percentage of patients who had SAC/VAL prescriptions rejected by an insurance payer | Up to 3 months

SECONDARY OUTCOMES:
Percentage of patients who utilized a heart failure-related treatment in the follow-up period | Up to 12 months
Time to first angiotensin-converting enzyme inhibitor (ACEi), angiotensin II receptor blockers (ARB), or angiotensin-receptor neprilysin inhibitors (ARNI, i.e., SAC/VAL) in the follow-up period | Up to 12 months
Percentage of patients who had a disruption in the use of ACEi/ARB/ARNI in the follow-up period | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- IQVIA, Durham, North Carolina, United States